CLINICAL TRIAL: NCT05375890
Title: Clinical and Neurophysiological Characteristics of Narcolepsy in Russia Basing on Clinical, Polysomnographic and Genome-wide Association Analyses of Narcolepsy With Cataplexy: a European Narcolepsy Network Study of 2013
Brief Title: Clinical and Neurophysiological Characteristics of Narcolepsy
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 246188
Record Dates: First submitted 2022-05-04; First posted 2022-05-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2022-05

CONDITIONS: Narcolepsy Type 1
Keywords: narcolepsy; cataplexy; excessive sleepiness; PSG; MSLT; Russia
MeSH Terms: conditions — Narcolepsy; Cataplexy; Disorders of Excessive Somnolence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — Narcolepsy patients in Russia gathered according to criteria.

SUMMARY:
The study is the first attempt in post-Soviet Russian history to collect and analyze the existing available data of narcolepsy cohort in order to get prove characteristics of narcolepsy in Russia according to known data. Investigators created the system of national narcolepsy centers in Russia - Russian narcolepsy network, with a purpose of collecting clinical and neurophysiological data with subsequent analyze and formation of Russian narcolepsy profile.

DETAILED DESCRIPTION:
First reports of narcolepsy with cataplexy in Russia were made by Mankovsky in 1925 (narcolepsy with cataplexy, NC). The largest series of patients (n=110) was reported by A. Vein in 1964. Narcolepsy remains however until today relatively unknown in Russia. The aim of this study is to report clinical and polysomnographic (PSG)/multiple sleep latency test (MSLT) results in a Russian population and compare them with the European narcolepsy network (n=1099) reported (Luca G, Haba-Rubio J, Dauvilliers Y, Lammers GJ, Overeem S, Donjacour CE, Mayer G, Javidi S, Iranzo A, Santamaria J, Peraita-Adrados R, Hor H, Kutalik Z, Plazzi G, Poli F, Pizza F, Arnulf I, Lecendreux M, Bassetti C, Mathis J, Heinzer R, Jennum P, Knudsen S, Geisler P, Wierzbicka A, Feketeova E, Pfister C, Khatami R, Baumann C, Tafti M; European Narcolepsy Network. Clinical, polysomnographic and genome-wide association analyses of narcolepsy with cataplexy: a European Narcolepsy Network study. J Sleep Res. 2013 Oct;22(5):482-95. doi: 10.1111/jsr.12044. Epub 2013 Mar 18. PMID: 23496005., 2013).

For the purpose of this study only patients with narcolepsy with cataplexy were considered because of the uncertainty about the diagnosis of narcolepsy without cataplexy.

In order to create a network of sleep centers with expertise/interest in narcolepsy 79 centers from 27 Russian cities were connected in 2019. A total of 11 centers officially joined the Russian Narcolepsy Network (rnane.ru) and agreed to participate in the current study. A standardized questionnaire, similar to the one reported by the EU-NN in a series of 1099 patients (Luca G, Haba-Rubio J, Dauvilliers Y, Lammers GJ, Overeem S, Donjacour CE, Mayer G, Javidi S, Iranzo A, Santamaria J, Peraita-Adrados R, Hor H, Kutalik Z, Plazzi G, Poli F, Pizza F, Arnulf I, Lecendreux M, Bassetti C, Mathis J, Heinzer R, Jennum P, Knudsen S, Geisler P, Wierzbicka A, Feketeova E, Pfister C, Khatami R, Baumann C, Tafti M; European Narcolepsy Network. Clinical, polysomnographic and genome-wide association analyses of narcolepsy with cataplexy: a European Narcolepsy Network study. J Sleep Res. 2013 Oct;22(5):482-95. doi: 10.1111/jsr.12044. Epub 2013 Mar 18. PMID: 23496005., 2013) was sent by mail to the 11 centers. The questionnaire included the following parameters:

1. Demographic characteristics: date of birth, gender, height, weight, BMI(body mass index) at diagnosis.
2. Age at EDS (excessive daytime sleepines) onset and age at cataplexy onset. Investigators defined the age at onset of NC(narcolepsy with cataplexy) as the age at occurrence of EDS and/or cataplexy, determined during the clinical interview.
3. Frequency of cataplexy attacks at diagnosis. The frequency of cataplexy was assessed by a scale from 1 to 5, reporting rare to very frequent cataplexy attacks: 1 = one or less cataplexy attacks per year; 2 = more than one cataplexy attack per year but less than one per month; 3 = more than one attack per month but less than one per week; 4 = more than one per week but less than one per day; 5 = at least one cataplexy attack per day.
4. ESS (Epworth Sleepiness Scale) score at diagnosis.
5. Polysomnographic variables [sleep onset latency at diagnosis, apnea-hypopnea index (AHI) and periodic leg movements during sleep index (PLMSI) when available] and MSLT results (mean sleep latency, number of SOREMPs) at diagnosis. Even if the recording procedures were different among centers, most of the patients underwent nocturnal in-lab PSG followed by an MSLT as part of the diagnostic evaluation. For PSG and MSLT, sleep latency was defined as the time from lights off to the first epoch scored as sleep. A SOREMP was defined as the occurrence of an epoch of REM(rapid eye movement) sleep within 15 min after the first epoch scored as sleep. Although MSLT was performed according to standard methods (Carskadon MA, Dement WC, Mitler MM, Roth T, Westbrook PR, Keenan S. Guidelines for the multiple sleep latency test (MSLT): a standard measure of sleepiness. Sleep. 1986 Dec;9(4):519-24. doi: 10.1093/sleep/9.4.519. PMID: 3809866.), the number of scheduled naps could be variable. To standardize the results, investigators calculated the percentage of SOREMPs of the total number of naps: percentage of naps with SOREMPs.

7. Associated features, with particular attention to symptoms frequently reported with narcolepsy: sleep paralysis (SP); hypnagogic/hypnopompic hallucinations (HH); and poor nocturnal sleep.

8. Co-morbidities (sleep-related, somatic or psychiatric) and treatment when available.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent of the patient and/or parent/adoptive parent (in the case of a minor) to participate in the study;
2. Age: 6-80 years;
3. Gender: Men and women;
4. Established diagnosis: Narcolepsy of type I and II (according to the criteria of the International classification of sleep disorders of 2014).

Exclusion Criteria:

1. Refusal of the patient or his parent / adoptive parent (in the case of a minor) from further participation in the study;
2. The occurrence of a serious illness or a significant deterioration of a disease unrelated to narcolepsy;
3. Pregnancy started after inclusion.

Ages: 7 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men and women aged 6-80 who have been diagnosed with narcolepsy type I, met inclusion criteria and who(or whose representatives in case of being under 18 years) agreed to participate in studying.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
date of birth | during 1-3 years after beginning and when patient and data are available
  year of birth
gender | during 1-3 years after beginning and when patient and data are available
  male or female
height | during 1-3 years after beginning and when patient and data are available
  meters
weight | during 1-3 years after beginning and when patient and data are available
  kilograms
BMI at diagnosis | during 1-3 years after beginning and when patient and data are available
  Weight and height will be combined to report BMI in kg/m^2 at the time of diagnosis
age at EDS (excessive daytime sleepioness) onset | during 1-3 years after beginning and when patient and data are available
  Age when EDS first time was reported by patient
age at cataplexy onset | during 1-3 years after beginning and when patient and data are available
  Age when cataplexy first time was reported by patient
frequency of cataplexy attacks at diagnosis | during 1-3 years after beginning and when patient and data are available
  Reported at diagnosis. The frequency of cataplexy was assessed by a scale from 1 to 5, reporting rare to very frequent cataplexy attacks: 1 = one or less cataplexy attacks per year; 2 = more than one cataplexy attack per year but less than one per month; 3 = more than one attack per month but less than one per week; 4 = more than one per week but less than one per day; 5 = at least one cataplexy attack per day.
ESS score at diagnosis | during 1-3 years after beginning and when patient and data are available
  Unit of Measure at diagnosis
Apnea-hypopnea index (AHI) | during 1-3 years after beginning and when patient and data are available
  PSG at diagnosis, Unit of Measure at diagnosis
Periodic leg movements during sleep index (PLMSI) | during 1-3 years after beginning and when patient and data are available
  Number of episodes and hours of sleep combined to report PLMSI in episodes per hour.
Sleep onset latency at diagnosis | during 1-3 years after beginning and when patient and data are available
  Time from lights off to the first epoch scored as sleep in PSG. Measured in minutes.
Sleep latency | during 1-3 years after beginning and when patient and data are available
  Time from lights off to the first epoch scored as sleep in MSLT. Measured in minutes.
Number of SOREM | during 1-3 years after beginning and when patient and data are available
  It was defined as the occurrence of an epoch of REM sleep within 15 min after the first epoch scored as sleep. Then investigators calculated the percentage of SOREMPs of the total number of naps: percentage of naps with SOREMPs.
Frequently of sleep paralysis, hypnagogic/hypnopompic hallucinations and poor nocturnal sleep, co-morbidities (sleep-related, somatic or psychiatric) and treatment when available. | during 1-3 years after beginning and when patient and data are available
  Percentage of occurence in group.

SECONDARY OUTCOMES:
summarization of collected database with European one | 1 year after receiving data from sleep centers from Russia and publishing results
  analyzing and comparison collected data with European one leading to final summarization of studying

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kuts, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (11):
- Russia (11):
  - Regional Clinical Hospital No.3, Chelyabinsk
  - Kazan State Medical University, Kazan'
  - Private healthcare institution 'Clinical hospital 'RZD-Medicine', Khabarovsk
  - Burnasyan Federal Medical Biophysical Center of Federal Medical Biological Agency, Moscow
  - FSBI NMRCO FMBA Russia, Moscow
  - I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow
  - Novosibirsk State Medical University, Novosibirsk
  - Almazov National Medical Research Centre, Saint Petersburg
  - Nikiforov Russian Center of Emergency and Radiation Medicine, EMERCOM of Russia, Saint Petersburg
  - V. M. Bekhterev National Research Medical Center for Psychiatry and Neurology, Saint Petersburg
  - Samara State Medical University, Samara

IPD SHARING:
Plan to Share IPD: Yes
IPD Sharing can be done after written official request in Sechenov University and approval of Central Contact investigator because our local Ethics committee does not allow free study sharing.
Time Frame: After official request and approval the data will become available with an indication of the terms of use.
Access Criteria: Our Ethics committee does not approve free study sharing. We can provide it only after written official request in Sechenov University and approval of Central Contact investigator.

REFERENCES:
- [Background] Kuts A, Poluektov M, Bassetti CLA. The evolution of the narcolepsy concept in Russia: A historical view. J Hist Neurosci. 2021 Apr-Jun;30(2):113-127. doi: 10.1080/0964704X.2020.1777502. Epub 2020 Jun 30. PMID 32603636
- [Derived] Kuts A, Poluektov M, Zakharov A, Govzman V, Ponomareva I, Yakupov E, Zavalko I, Tikhomirova O, Sviryaev Y, Yakovlev A, Polyakov A, Melnikov A, Bassetti CLA. Clinical and neurophysiological characteristics of 89 patients with narcolepsy and cataplexy from the Russian Narcolepsy Network. J Clin Sleep Med. 2023 Feb 1;19(2):355-359. doi: 10.5664/jcsm.10340. PMID 36305577
- See also: Official website of Russian narcolepsy network — http://www.rnane.ru